CLINICAL TRIAL: NCT06344910
Title: PRagmatic Study Of Messaging to Providers of Patients With Heart Failure in Amsterdam UMC
Acronym: PROMPT-HF-AUMC
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: AstraZeneca (Industry); Yale University (Other)
Responsible Party: Principal Investigator, Prof. Dr. Folkert W. Asselbergs, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 20230416-C1_v2
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: electronic health records; electronic nudge; guideline directed medical therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with HFrEF
  Interventions: Other: Best practice alert for the notification of patients with HFrEF and recommended evidence-based therapies

INTERVENTIONS:
Other: Best practice alert for the notification of patients with HFrEF and recommended evidence-based therapies — An algorithm will check if the patients if the patient has an age >18 year and is treated at the cardiology department for HFrEF. The use of GDMT is determined using prescriptions data electronic health records (EHR). If the patient does not receive treatment for all 4 drug classes (ACE/ARB/ARNi, beta-blocker, MRA, SGLT2-inhibitor), an electronic alert will be displayed suggesting the clinician to prescribe additional medication when clinically indicated, including relevant recent laboratory results (renal function and electrolytes) and other relevant measures (LVEF, blood pressure and heart rate). The alert is linked to an order set to aid in the prescription of GDMT according to current guidelines.
  Results will compared to a retrospective cohort (t=-12 to t=-6) months, and a silent mode cohort (t=-6 to t=0 months, in which a paired and a before and after analysis will be performed to evaluate the effect of the alert.

SUMMARY:
This is a prospective cohort study, where the investigators aim to investigate the effect of implementation of an electronic nudge alerting clinicians to the prescription of the 4 key pharmacological classes for the treatment of patients with heart failure and reduced ejection fraction (HFrEF) at the outpatient clinic in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Treatment for HFrEF at the outpatient clinic cardiology.
* Documented reduced ejection fraction of <40% based on cardiac ultrasound or cardiac magnetic resonance imaging.

Exclusion Criteria:

* Opt-out for the use of routine clinical data for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with heart failure and reduced ejection fraction
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Use of guideline-directed medical therapy (GDMT) | 30 days (primary), 6 months (secondary)
  Using all therapies according to ESC guidelines

SECONDARY OUTCOMES:
All-cause mortality | 1 year
  All-cause mortality
Hospitalisation for Heart Failure | 6 months, 1 year
  Hospitalisation for Heart Failure
other major cardiovascular events (MACE: cardiovascular death, non-fatal myocardial infarction, non-fatal stroke) | 6 months, 1 year
  other major cardiovascular events (MACE: cardiovascular death, non-fatal myocardial infarction, non-fatal stroke)
renal events (>30% serum creatinine increase, hospitalization for acute kidney injury, development of end-stage kidney disease) | 30 days, 6 months, 1 year
  renal events (>30% serum creatinine increase, hospitalization for acute kidney injury, development of end-stage kidney disease)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam University Medical Centers, Location AMC, Amsterdam
  - Amsterdam University Medical Centers, Location VU Medical Center, Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data underlying the results for publication can be made available upon request
Supporting Information: Study Protocol, SAP
Time Frame: available upon request
Access Criteria: available upon request